CLINICAL TRIAL: NCT05338515
Title: A Phase I, Single-Ascending Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of LOXO-292 in Healthy Adult Subjects
Brief Title: A Study of Selpercatinib (LY3527723) in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Loxo Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 17485; J2G-OX-JZJF (Other: Eli Lilly and Company); LOXO-RET-18057 (Other: Loxo Oncology, Inc.)
Record Dates: First submitted 2022-04-19; First posted 2022-04-21 (Actual); Results first posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Healthy
MeSH Terms: interventions — selpercatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 320 mg Selpercatinib (Experimental): Participants received a single oral dose of 320 mg selpercatinib on Day 1, preceded by an overnight fast of at least 10 hours, followed by a fast from food (not including water) for at least 4 hours post dose.
  Interventions: Drug: Selpercatinib
- 640 mg Selpercatinib (Experimental): Participants received a single oral dose of 640 mg selpercatinib on Day 1, preceded by an overnight fast of at least 10 hours, followed by a fast from food (not including water) for at least 4 hours post dose.
  Interventions: Drug: Selpercatinib
- 720 mg Selpercatinib (Experimental): Participants received a single oral dose of 720 mg selpercatinib on Day 1, preceded by an overnight fast of at least 10 hours, followed by a fast from food (not including water) for at least 4 hours post dose.
  Interventions: Drug: Selpercatinib

INTERVENTIONS:
Drug: Selpercatinib — Administered orally.
  Other Names: LY3527723; LOXO-292

SUMMARY:
The main purpose of this study is to determine how safe and how well tolerated selpercatinib is when given as oral doses to healthy participants. The study will also assess how fast selpercatinib gets into the blood stream and how long it takes the body to remove it. The study will last up to about 6 weeks, inclusive of screening period.

ELIGIBILITY:
Inclusion Criteria:

* Female participants of non-childbearing potential who are agreeable to take birth control measures until study completion
* Body mass index (BMI) ≥ 18.0 and ≤ 32.0 kilograms per meter squared (kg/m²) and had a minimum weight of at least 50 kg at screening
* Have normal blood pressure, pulse rate, electrocardiogram (ECG), and blood and urine laboratory test results that are acceptable for the study

Exclusion Criteria:

* Are currently participating in or completed a clinical trial within the last 30 days or any other type of medical research judged to be incompatible with this study
* Have previously participated or withdrawn from this study
* Have or used to have health problems or laboratory test results or ECG readings that, in the opinion of the doctor, could make it unsafe to participate, or could interfere with understanding the results of the study
* Had blood loss of more than 500 milliliters (mL) within the previous 30 days of study screening
* Require treatment with inducers or inhibitors of cytochrome P450 (CYP) CYP3A within 14 days before the first dose of study drug through the end of Period 2

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2019-02-12 (Actual); Primary Completion 2019-03-12 (Actual); Study Completion 2019-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Celerion, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- 320 Milligram (mg) Selpercatinib: Participants received a single oral dose of 320 mg selpercatinib on Day 1, preceded by an overnight fast of at least 10 hours, followed by a fast from food (not including water) for at least 4 hours post dose.
Period: Overall Study
Arm/Group | 320 Milligram (mg) Selpercatinib | 640 mg Selpercatinib | 720 mg Selpercatinib
Started | 6 | 6 | 6
Received at Least One Dose of Study Drug | 6 | 6 | 6
Completed | 6 | 6 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | 320 mg Selpercatinib | 640 mg Selpercatinib | 720 mg Selpercatinib | Total
Number analyzed (Participants) | 6 | 6 | 6 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.8 (7.19) | 36.7 (10.69) | 39.3 (9.99) | 37.9 (8.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 3 | 5
  Male | 5 | 5 | 3 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 4 | 10
  Not Hispanic or Latino | 3 | 3 | 2 | 8
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 1 | 3
  White | 4 | 4 | 4 | 12
  More than one race | 1 | 1 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 6 | 6 | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration
Description: Data presented are the number of participants who experienced SAEs considered by the investigator to be related to study drug administration. A summary of SAEs and all other non-serious Adverse Event(s) (AEs), regardless of causality, is located in the Reported Adverse Event module.
Time Frame: Baseline up to Day 8
Population: All randomized participants who received at least one dose of study drug and had at least one post dose safety assessment.
Measure: Number; unit: participants
Arm/Group | 320 mg Selpercatinib | 640 mg Selpercatinib | 720 mg Selpercatinib
Number analyzed (Participants) | 6 | 6 | 6
participants | 0 | 0 | 0

2. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration-time Curve, From Time 0 to the Last Observed Non-zero Concentration (AUC0-t) of Selpercatinib
Description: PK: AUC0-t is calculated using the linear trapezoidal with linear interpolation method.
Time Frame: Predose (within 30 minutes), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144 and 168 hours postdose
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*h/ mL)
Arm/Group | 320 mg Selpercatinib | 640 mg Selpercatinib | 720 mg Selpercatinib
Number analyzed (Participants) | 6 | 6 | 6
nanogram*hour per milliliter (ng*h/ mL) | 35900 (59.7) | 50460 (46.5) | 60960 (50.7)

3. Secondary Outcome: PK: Area Under the Concentration-time Curve, From Time 0 to Hour 24 (AUC0-24) of Selpercatinib
Description: PK: AUC0-24 was calculated using the linear trapezoidal with linear interpolation method.
Time Frame: Predose (within 30 minutes), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 hours postdose
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/ mL
Arm/Group | 320 mg Selpercatinib | 640 mg Selpercatinib | 720 mg Selpercatinib
Number analyzed (Participants) | 6 | 6 | 6
ng*h/ mL | 21280 (79.8) | 30680 (50.5) | 36450 (58.3)

4. Secondary Outcome: PK: Area Under the Concentration-time Curve From Time 0 Extrapolated to Infinity (AUC0-inf) of Selpercatinib
Description: PK: AUC0-inf was calculated as AUC0-inf = AUC0-t + (Clast/Kel) where Clast is the last observed/measured concentration and Kel is the apparent terminal elimination rate constant, which represents the fraction of drug eliminated per unit time.
Time Frame: as for outcome 2
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*h/ mL)
Arm/Group | 320 mg Selpercatinib | 640 mg Selpercatinib | 720 mg Selpercatinib
Number analyzed (Participants) | 6 | 6 | 6
nanogram*hour per milliliter (ng*h/ mL) | 36080 (59.7) | 50770 (46.7) | 61380 (50.7)

5. Secondary Outcome: PK: Percent of AUC0-inf Extrapolated (AUC%Extrap) of Selpercatinib
Description: PK: Percent of AUC0-inf extrapolated was calculated as (1-AUC0-t/AUC0-inf) *100.
Time Frame: Predose -168 hours post dose
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | 320 mg Selpercatinib | 640 mg Selpercatinib | 720 mg Selpercatinib
Number analyzed (Participants) | 6 | 6 | 6
percentage | 0.5159 (0.44688) | 0.6238 (0.29008) | 0.6869 (0.29427)

6. Secondary Outcome: PK: Apparent Total Plasma Clearance After Oral (Extravascular) Administration (CL/F) of Selpercatinib
Description: PK: CL/F was calculated as Dose/(AUC0-inf).
Time Frame: as for outcome 2
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data.
Measure: Mean (Standard Deviation); unit: Liters per Hour (L/h)
Arm/Group | 320 mg Selpercatinib | 640 mg Selpercatinib | 720 mg Selpercatinib
Number analyzed (Participants) | 6 | 6 | 6
Liters per Hour (L/h) | 10.16 (6.3442) | 13.62 (5.5060) | 12.79 (5.2828)

7. Secondary Outcome: PK: Maximum Observed Concentration (Cmax) of Selpercatinib
Description: PK: Cmax was taken directly from bioanalytical data.
Time Frame: as for outcome 2
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | 320 mg Selpercatinib | 640 mg Selpercatinib | 720 mg Selpercatinib
Number analyzed (Participants) | 6 | 6 | 6
nanograms per milliliter (ng/mL) | 2282 (88.6) | 3316 (56.3) | 3745 (55.2)

8. Secondary Outcome: PK: Time to Reach Cmax (Tmax) of Selpercatinib
Description: PK: Tmax was time to reach Cmax. If the maximum value occurs at more than one time point, Tmax is defined as the first time point with this value taken from clinical database as the difference in the time of administration and the time of the blood draw which is associated with the Cmax.
Time Frame: as for outcome 2
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data.
Measure: Median (Full Range); unit: hour
Arm/Group | 320 mg Selpercatinib | 640 mg Selpercatinib | 720 mg Selpercatinib
Number analyzed (Participants) | 6 | 6 | 6
hour | 2.001 [1.50 to 3.00] | 1.999 [1.03 to 2.51] | 2.753 [2.00 to 4.00]

9. Secondary Outcome: PK: Apparent First-order Terminal Elimination Rate Constant (Kel) of Selpercatinib
Description: PK: Apparent terminal elimination rate constant; represents the fraction of drug eliminated per unit time calculated by linear least squares regression analysis using the maximum number of points in the terminal log linear phase (e.g., three or more non zero plasma concentrations).
Time Frame: as for outcome 2
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data.
Measure: Mean (Standard Deviation); unit: 1/hour (1/h)
Arm/Group | 320 mg Selpercatinib | 640 mg Selpercatinib | 720 mg Selpercatinib
Number analyzed (Participants) | 6 | 6 | 6
1/hour (1/h) | 0.03122 (0.0094408) | 0.02607 (0.0054791) | 0.02562 (0.0040999)

10. Secondary Outcome: PK: Apparent Volume of Distribution During the Terminal Elimination Phase (Vz/F) of Selpercatinib
Description: PK: Vz/F calculated as Dose/(AUC0-inf x Kel).
Time Frame: as for outcome 2
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data.
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | 320 mg Selpercatinib | 640 mg Selpercatinib | 720 mg Selpercatinib
Number analyzed (Participants) | 6 | 6 | 6
Liter | 328.7 (156.37) | 526.3 (219.99) | 487.0 (158.59)

ADVERSE EVENTS:
Time Frame: Baseline up to Day 8
Description: All randomized participants who received at least one dose of study drug.
Arm/Group | 320 mg Selpercatinib | 640 mg Selpercatinib | 720 mg Selpercatinib
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 1/6 | 1/6 | 4/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 320 mg Selpercatinib (N=6) | 640 mg Selpercatinib (N=6) | 720 mg Selpercatinib (N=6)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Ulcer (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Burning sensation (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Papule (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-01-25): https://cdn.clinicaltrials.gov/large-docs/15/NCT05338515/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-03): https://cdn.clinicaltrials.gov/large-docs/15/NCT05338515/SAP_001.pdf